CLINICAL TRIAL: NCT01464970
Title: The Potential Role of the Superficial Inferior Epigastric Vascular System in the Perfusion of Zone IV of Deep Inferior Epigastric Perforator (DIEP) Flaps
Brief Title: Influence of the Superficial Inferior Epigastric System in Deep Inferior Epigastric Perforator (DIEP) Flaps
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: Canniesburn Research Trust (Unknown)
Responsible Party: Principal Investigator, Adam Gilmour, Principal Investigator - Clinical Laser Research Fellow, NHS Greater Glasgow and Clyde
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: GN11CA415
Record Dates: First submitted 2011-10-30; First posted 2011-11-04 (Estimated); Last update posted 2012-05-14 (Estimated); Status verified 2012-05

CONDITIONS: Breast Cancer
Keywords: DIEP perfusion; Zone IV; Free Flap; Breast Cancer Reconstruction; Perfusion of Zone IV of DIEP flaps
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- SIE Vessels Both Clamped (Active Comparator)
  Interventions: Procedure: Both Superficial Inferior Artery and Vein Clamped
- SIE Vessels both Unclamped (Active Comparator)
  Interventions: Procedure: Superficial Inferior Epigastric Vessels both unclamped
- SIE Artery Unclamped; Vein Clamped (Active Comparator)
  Interventions: Procedure: SIE Artery Unclamped, Vein Clamped
- SIE Artery Clamped, SIE Vein Unclamped (Active Comparator): Superficial Inferior Epigastric Artery Clamped; Vein Unclamped
  Interventions: Procedure: SIE Artery clamped, Vein unclamped

INTERVENTIONS:
Procedure: Both Superficial Inferior Artery and Vein Clamped — Perfusion assessed in Zone IV of the DIEP flap whilst both the contralateral Superficial Inferior Epigastric Artery and Vein are clamped
  Arms: SIE Vessels Both Clamped
Procedure: Superficial Inferior Epigastric Vessels both unclamped — Perfusion assessed in Zone IV of the DIEP flap whilst both the contralateral Superficial Inferior Epigastric Artery and Vein are unclamped
  Arms: SIE Vessels both Unclamped
Procedure: SIE Artery Unclamped, Vein Clamped — Perfusion assessed in Zone IV of the DIEP flap whilst the contralateral Superficial Inferior Epigastric Artery is unclamped and the Vein is clamped
  Arms: SIE Artery Unclamped; Vein Clamped
Procedure: SIE Artery clamped, Vein unclamped — Perfusion assessed in Zone IV of the DIEP flap whilst the contralateral Superficial Inferior Epigastric Artery is clamped and the Vein is unclamped
  Arms: SIE Artery Clamped, SIE Vein Unclamped

SUMMARY:
The purpose of this study is to determine in-vivo the effects the contralateral superficial inferior epigastric vascular system has on the perfusion of Zone IV of deep inferior epigastric perforator flaps.

DETAILED DESCRIPTION:
* Breast cancer is the commonest cancer to affect women in the UK. Current guidelines state that; disease permitting, all females due to undergo mastectomy for breast cancer should be offered reconstruction. Autologous free tissue transfer using abdominal tissue remains an excellent option for breast reconstruction due the readily available fatty tissue and the low donor site morbidity. In recent years the trend has been to base the abdominal tissue on perforating vessels rather than to routinely harvest muscle along with the flap; thus further potentially reducing donor site morbidity. Abdominal tissue based upon the Deep Inferior Epigastric Perforator (DIEP) system is a well recognised option in breast reconstruction.
* This procedure involves harvesting the lower abdominal tissue basing its blood supply on one of the Deep Inferior Epigastric Perforating Arteries and concomitant veins. These are branches of the External iliac artery which perforate through the rectus muscle or the intertendinous intersections.
* A large volume of tissue can be harvested based on a single perforator.
* Hartrampf divided the abdominal tissues into distinct perfusion zones I-IV based upon their location to the perforating artery. Zone I overlies the perforating vessel, Zone II is across the midline adjacent to perforating vessel. Zone III is on the ipsilateral periphery to the perforating vessel and Zone IV is on the furthest periphery on the contralateral side from the perforator. Over the years this has undergone debate and many have advocated that zones II-III (according to Hartrampfs original classification) should be switched. However everyone remains clear on the term Zone IV. Zone IV is classically the area of the flap which receives least perfusion/drainage from the perforating vessels and as such is most liable to undergo congestion and tissue ischaemia leading to fat/skin necrosis. As such many surgeons routinely excise zone IV from the DIEP flap prior to transfer to the chest defect. This obviously leads to a reduction in the volume of tissue available for reconstruction.
* Classically most problems with zone IV / flap perfusion tend to be related to venous congestion.
* Many surgeons advocate the use of the superficial inferior epigastric vein as a "lifeboat" vessel in salvaging a congested DIEP and have published their results in doing so.
* There are however no in-vivo studies showing the full contribution of the superficial vascular system in flaps based primarily upon the Deep Inferior Epigastric Perforating Vessels. A recent study using preoperative CTs has shown that there are "macrovascular-shunts" between the deep arterial system and the superficial venous system but the implications of this have yet to be established.
* Fluoroscopy using indocyanine green is an established method at looking at tissue perfusion in free flaps.
* Laser Doppler imaging is another well described technique for the monitoring / assessment of tissue perfusion in plastic surgery operations.
* By further understanding the perfusion of the DIEP flaps the investigators hope to improve flap survivability and also the volume of flap which can be used.
* Patients due to undergo breast reconstruction with a free DIEP flap by the senior researcher/surgeon will be identified.
* On the day of their operation the DIEP flap will be raised as normal on one of the DIEP arteries from either side. The superficial vascular system will be dissected free on the contralateral side.
* The flap will then be scanned with Laser Doppler Imaging and then the SPY scanner (indocyanine green angiography coupled with fluoroscopy)
* This will take place in a randomized fashion as follows
* Superficial Inferior Epigastric Artery Clamped; Vein Unclamped
* Superficial Inferior Epigastric Artery Unclamped; Vein Clamped
* Both Artery and Vein Clamped
* Both Artery And Vein Unclamped
* There will be a 5minute pause between each intervention to allow perfusion to stabilize. Previous research (awaiting publication) within our department has shown that this is the necessary amount of time to allow stabilization.
* The scanning period will be carried out during the natural rest break of the operating surgeon and as such will not add significantly to the length of the procedure.
* Once the scanning process is finished the operation will then proceed as standard with DIEP flap being disconnected from the abdomen and reconnected in the chest to reconstruct the breast.

ELIGIBILITY:
Inclusion Criteria:

* Female Patient
* Ages 18-70 years old
* Undergoing unilateral DIEP flap reconstruction post mastectomy.

Exclusion Criteria:

* Hyperthyroidism / history of autonomic thyroid adenoma (slightly increased risk of allergic reaction to the dye)
* ASA grade 3+
* Abdominal Scarring

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2011-12; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Deep Inferior Epigastric Perforator Flap Zone IV Tissue Perfusion | Intra-Operatively
  Tissue Perfusion to Zone IV will be assessed intra-operatively using Laser Doppler Imaging and angiography whilst various components of the Contralateral Superficial Inferior Epigastic Artery / Vein are clamped/unclamped.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Gilmour, MBChB, MRCS (Ed), Principal Investigator — Canniesburn Plastic Surgery Unit
Locations (1):
- Canniesburn Plastic Surgery Unit, Glasgow Royal Infirmary, Glasgow, United Kingdom